CLINICAL TRIAL: NCT01378910
Title: Use Of Genotypic HIV-1 Tropism Testing In Proviral DNA To Guide CCR5 Antagonist Treatment In Subjects With Undetectable HIV-1 Viremia
Brief Title: Genotypic Tropism Testing In Proviral Dna To Guide CCR5 Antagonist Treatment In Subjects With Undetectable HIV-1 Viremia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PROTEST
Record Dates: First submitted 2011-06-17; First posted 2011-06-23 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2014-07

CONDITIONS: HIV
Keywords: HIV; TROPISM; PBMC; GENOTYPE; 454 SEQUENCING

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Change of 3rd drug to maraviroc (Experimental): Change of PI, NNRTI or integrase inhibitor to CCR5 antagonist (maraviroc)
  Interventions: Drug: Unique

INTERVENTIONS:
Drug: Unique — Change of PI, NNRTI or integrase inhibitor to CCR5 antagonist (maraviroc)

SUMMARY:
CCR5 antagonists might be an adequate alternative for HIV-1-infected individuals with suppressed viremia who experience antiretroviral-related toxicity. The assessment of HIV-1 tropism in proviral DNA could be helpful to inform in which of these subjects CCR5 antagonists could be efficacious.

DETAILED DESCRIPTION:
The assessment of HIV-1 tropism is needed before starting treatment with a CCR5-antagonist. Several phenotypic and genotyping tropism tests have been developed in the recent years. Phenotypic assays (i.e. TrofileTM and ES-TrofileTM) have been used.in most clinical trials. Genotypic tropism testing, however, is easier, cheaper and faster than phenotypic methods, and can be performed in a local HIV laboratories.

Viral RNA amplification is difficult in subjects with HIV-1 RNA levels <500-1000 copies/mL. In these cases, the optimal source of genetic material is peripheral blood mononuclear cell (PBMC)-associated proviral DNA. Whereas genotypic tropism testing in proviral DNA is technically feasible, it has not been validated as a tool to predict sustained virological response to CCR5-antagonist therapy in subjects with undetectable viremia.

As of today, maraviroc is the only CCR5-antagonist approved for HIV treatment. It has few drug interactions and a good security profile, particularly in terms of lipid and glucose metabolism. Therefore, it might be an adequate alternative for HIV-1-infected individuals with suppressed viremia who experience antiretroviral-related toxicity or metabolic problems.

This study will evaluate 48-week virological outcomes in aviremic subjects with an R5 virus by proviral genotypic tropism testing who switch the "third drug" of their regimen to maraviroc.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected patients.
2. Age 18 or more.
3. Antiretroviral treatment containing 2 Nucleoside/Nucleotide Reverse Transcriptase Inhibitors (NRTIs) plus 1 Non-nucleoside reverse-transcriptase inhibitor (NNRTI) or 1 protease inhibitor (PI) or 1 integrase inhibitor (ININ)
4. Patients receiving stable antiretroviral treatment for at least 6 months.
5. Viral load under 50 copies/mL in the last 6 months
6. Patients with CCR5 tropism based in V3 genotyping in proviral DNA using the G2P with a false positive rate of 10% interpretation method.
7. A change of treatment is needed due to toxicity / tolerability problems with the 3rd drug (PI, NNRTI or ININ), according to investigator criteria.
8. An antiretroviral regimen containing a CCR5-antagonist is suitable for the patient (physician criteria).
9. Voluntary written informed consent.

Exclusion Criteria:

1. Pregnancy or breast-feeding.
2. Patient previously treated with maraviroc.
3. Patients with documented resistance to maraviroc or any other drug considered for the new ARV regimen.
4. Viral failure in the moment of inclusion.
5. Bad adherence history or anticipated (investigator criteria).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-06; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with viral load under 50 copies/mL | Week 48

SECONDARY OUTCOMES:
Percentage of patients without confirmed virological failure. | Up to week 48
  To evaluate other aspects related to maintanence of virological response.
Time to loss of virological response (TLOVR) < 200 copies/mL | Up to week 48
  To evaluate other aspects related to maintanence of virological response.
Time to loss of virological response (TLOVR) < 50 copies/mL | Up to week 48
  To evaluate other aspects related to maintanence of virological response.
Proportion of patients treated with maraviroc with viral load under 50 copies/mL | Week 12
  To evaluate other aspects related to maintanence of virological response
Proportion of patients treated with maraviroc with viral load under 50 copies/mL | Week 24
  To evaluate other aspects related to maintanence of virological response
Proportion of patients treated with maraviroc with viral load under 50 copies/mL | Week 36
  To evaluate other aspects related to maintanence of virological response
Proportion of patients treated with maraviroc with viral load under 50 copies/mL | Week 48
  To evaluate other aspects related to maintanence of virological response.
Time to treatment discontinuation, overall, and due to factors other than loss of virological response | Up to week 48
  To evaluate other aspects related to maintanence of virological response
Association between pre-treatment level of X4 viruses detected by deep sequencing at screening and virological response to maraviroc based therapy at week 48. | Week 48
  To evaluate changes in HIV tropism
Level of X4 viruses by detected by population sequencing. | Screening (up to 48 weeks)
  Evolution of viral tropism in PBMC-associated DNA by population and deep sequencing between screening and week 48 in subjects treated with maraviroc.
Level of X4 viruses by detected by population sequencing. | Week 12
  Evolution of viral tropism in PBMC-associated DNA by population and deep sequencing between screening and week 48 in subjects treated with maraviroc.
Level of X4 viruses by detected by population sequencing. | Week 48
  Evolution of viral tropism in PBMC-associated DNA by population and deep sequencing between screening and week 48 in subjects treated with maraviroc.
Level of X4 viruses by detected by deep sequencing. | Screening (up to 48 weeks)
  Evolution of viral tropism in PBMC-associated DNA by population and deep sequencing between screening and week 48 in subjects treated with maraviroc.
Level of X4 viruses by detected by deep sequencing. | Week 12
  Evolution of viral tropism in PBMC-associated DNA by population and deep sequencing between screening and week 48 in subjects treated with maraviroc.
Level of X4 viruses by detected by deep sequencing. | Week 48
  Evolution of viral tropism in PBMC-associated DNA by population and deep sequencing between screening and week 48 in subjects treated with maraviroc.
High-resolution assessment of virus diversity and X4 level using deep sequencing | Week 12
  High-resolution assessment of virus diversity and X4 level using deep sequencing at week 12 and at the time of virological failure.
High-resolution assessment of virus diversity and X4 level using deep sequencing | In case of virological failure (week 12 up to virological failure)
  High-resolution assessment of virus diversity and X4 level using deep sequencing at week 12 and at the time of virological failure.
Median change of total cholesterol. | From baseline to week 48.
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Median change of HDL cholesterol. | From Baseline to week 48.
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Median change of LDL cholesterol. | From Baseline to week 48.
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Median change of triglycerides | From Baseline to week 48.
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Median change of AST serum levels. | From Baseline to week 48.
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Median change of ALT serum levels. | From Baseline to week 48.
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Median change of alkaline phosphatase serum levels. | From Baseline to week 48.
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Median change of total bilirubin serum levels. | From Baseline to week 48.
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Cumulative number of adverse events | Week 4
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Cumulative number of adverse events | Week 12
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Cumulative number of adverse events | Week 24
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Cumulative number of adverse events | Week 36
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Cumulative number of adverse events | Week 48
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Cumulative number of grade 3-4 adverse events | Week 4
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Cumulative number of grade 3-4 adverse events | Week 12
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Cumulative number of grade 3-4 adverse events | Week 24
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Cumulative number of grade 3-4 adverse events | Week 36
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Cumulative number of grade 3-4 adverse events | Week 48
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen
Proportion of patients withdrawn from the study and reason for study withdrawal | Up to week 48
  To evaluate the tolerability and safety with CCR5 antagonist containing regimen

CONTACTS AND LOCATIONS:
Locations (24):
- Spain (24):
  - Hospital Xeral de Vigo, Santiago de Compostela, A Coruña
  - Hospital de Elche, Elche, Alicante
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - H. U. Germans Trias i Pujol, Badalona, Barcelona
  - H. de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital U. Marqués de Valdecilla, Santander, Cantabria
  - Hospital General de Castellón, Castellon, Castelló
  - Hospital Sta. Lucía/ H. Sta. Mª del Rosell, Cartagena, Murcia
  - Hospital de Cruces, Bilbao, Vizcaya
  - Hospital Gral. U. de Alicante, Alicante
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de Mataró, Barcelona
  - Hospital Virgen de las Nieves, Granada
  - Hospital U. San Cecilio, Granada
  - Hospital U. Gregorio Marañón, Madrid
  - Hospital Carlos III, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Reina Sofía de Murcia, Murcia
  - Hospital Sant Pau i Santa Tecla, Tarragona
  - Hospital La Fe, Valencia
  - Hospital Gral. U. de Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - Hospital U. Dr. Peset, Valencia